CLINICAL TRIAL: NCT06839664
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅲ Clinical Study to Evaluate the Efficacy and Safety of HS-20094 in Overweight and Obese Subjects
Brief Title: A Study of HS-20094 in Chinese Adults with Overweight or Obesity
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20094-301
Record Dates: First submitted 2025-02-18; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- HS-20094 5mg (Experimental)
  Interventions: Drug: HS-20094 injection
- HS-20094 10mg (Experimental)
  Interventions: Drug: HS-20094 injection
- HS-20094 15mg (Experimental)
  Interventions: Drug: HS-20094 injection
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo injection

INTERVENTIONS:
Drug: HS-20094 injection — Administered SC
  Arms: HS-20094 10mg; HS-20094 15mg; HS-20094 5mg
Drug: Placebo injection — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to assess the Efficacy and safety of HS-20094 in overweight and obese patients. The study will last up to approximately 52 weeks.

DETAILED DESCRIPTION:
This is a phase Ⅲ, double-blind, randomised, placebo-controlled trial to assess the efficacy of HS-20094 in Chinese subjects with overweight or obesity. We enrolled adults (aged 18-65 years, both inclusive) with overweight (body-mass index [BMI] ≥24 kg/m2) accompanied by at least one obesity-related comorbidity or obesity (BMI ≥28 kg/m2) in China. Eligible participants were randomly assigned to receive once-weekly subcutaneous HS-20094 or placebo for 48 weeks. The co-primary endpoints were the percent change in bodyweight from baseline and the proportion of patients achieving weight loss≥5% from baseline after 48 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1.Male or female 18 to 65 years of age at the time of consent(cutoff value included).

  2. Body mass Index(BMI)≥28 kilograms per square meter(kg/m2),or ≥24 kg/m2 and previous diagnosis with at least one of the following comorbidities: prediabetes, hypertension, dyslipidemia, non-alcoholic fatty liver disease, obstructive sleep apnea.

  3. Weight change ≤5.0% after diet and exercise control for at least 12 weeks before screening.

Exclusion Criteria:

* 1. Diabetes mellitus 2. Weight change >5.0% after diet and exercise control for at least 12 weeks before screening 3. Have used or are currently using weight loss drugs within 3 months before screening 4. History of pancreatitis 5. Family or personal history of medullary thyroid carcinoma(MTC)or multiple endocrine neoplasia syndrome type 2(MEN-2) 6. History of moderate to severe depression, or have a history of serious mental illness 7. Any lifetime history of a suicide attempt 8. Have a history of significant atopy (severe allergic manifestations), multiple or severe drug allergies, or severe posttreatment hypersensitivity reactions 9. Have a history of any malignancy within the past 5 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, week 48
  Percent Change from Baseline in Body Weight
Percentage of Participants Who Achieve weight loss≥ 5% from Baseline | Baseline, week 48
  Percentage of Participants Who Achieve weight loss≥ 5% from Baseline

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve weight loss≥10% and 15% from Baseline | Baseline, week 4
  Percentage of Participants Who Achieve weight loss≥10% and 15% from Baseline
Change in waist circumference from baseline at week 48 | Baseline, week 48
  Change in waist circumference from baseline at week 48
Percentage change in body weight from baseline at week 24 | Baseline, week 24
  Percentage change in body weight from baseline at week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China